CLINICAL TRIAL: NCT04941755
Title: A Phase 1 Open-label, 2-Period Crossover Study to Assess the Effect of Acid-reducing Agent Famotidine on the Pharmacokinetics of BMS-986256 in Healthy Participants
Brief Title: A Study to Determine the Effect of Famotidine on the Drug Levels of BMS-986256 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IM026-029
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; BMS-986256; Famotidine; Gastric pH
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental)
  Interventions: Drug: BMS-986256; Drug: Famotidine
- Sequence BA (Experimental)
  Interventions: Drug: BMS-986256; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986256 — Specified dose on specified days
Drug: Famotidine — Specified dose on specified days
  Other Names: Pepcid

SUMMARY:
The purpose of this study is to investigate the effect of gastric pH changes induced by famotidine on the drug levels of BMS-986256.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, defined as having no clinically significant deviations from normal in medical history
* Weight ≥ 50 kg and body mass index between 18.0 kg/m2 and 32.0 kg/m2, inclusive, at screening
* Normal renal function at screening

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent gastrointestinal (GI) disease that could impact upon the absorption of study treatment
* Any major surgery within 4 weeks of study treatment administration
* Significant history of GI abnormalities

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986256 | Up to 19 days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) of BMS-986256 | Up to 19 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-986256 | Up to 19 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 45 days
Incidence of Serious Adverse Events (SAEs) | Up to 45 days
Incidence of clinically significant changes in clinical laboratory values: Hematology tests | Up to 45 days
Incidence of clinically significant changes in clinical laboratory values: Chemistry tests | Up to 45 days
Incidence of clinically significant changes in clinical laboratory values: Urinalysis tests | Up to 45 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 45 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 45 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 45 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 45 days
Incidence of clinically significant changes in Electrocardiogram (ECG) parameters: PR interval | Up to 45 days
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in ECG parameters: QRS | Up to 45 days
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Incidence of clinically significant changes in ECG parameters: QT interval | Up to 45 days
  The QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in ECG parameters: QTcF | Up to 45 days
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave
Ratio of Cmax of BMS-986256 (with famotidine versus without famotidine) | Up to 45 days
Ratio of AUC(0-T) of BMS-986256 (with famotidine versus without famotidine) | Up to 45 days
Ratio of AUC(INF) of BMS-986256 (with famotidine versus without famotidine) | Up to 45 days
Time of maximum observed plasma concentration (Tmax) of BMS-986256 | Up to 45 days
Apparent terminal plasma half-life (T-HALF) of BMS-986256 | Up to 45 days
Apparent total body clearance (CLT/F) of BMS-986256 | Up to 45 days
Apparent volume of distribution of terminal phase (Vz/F) of BMS-986256 | Up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm